CLINICAL TRIAL: NCT01694797
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-period, Two Sequence, Single Dose, Crossover, Oral Bioequivalence Study of Metoprolol Succinate Extended-Release Tablets 50 mg of Dr. Reddy's Laboratories Limited, India Comparing With That of TOPROL-XL® (Containing Metoprolol Succinate) Extended-Release Tablets 50 mg of AstraZeneca LP Wilmington, DE in Healthy, Adult, Human Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study for Metoprolol Succinate ER Tablets 50 mg Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 642/09
Record Dates: First submitted 2012-09-24; First posted 2012-09-27 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2010-11

CONDITIONS: Healthy
MeSH Terms: interventions — Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metoprolol Succinate ER Tablets, 50 mg (Experimental): Metoprolol Succinate ER Tablets, 50 mg of Dr.Reddy's Laboratories Ltd
  Interventions: Drug: Metoprolol Succinate
- TOPROL-XL ER Tablets 50 mg (Active Comparator): TOPROL-XL ER Tablets 50 mg of AstraZeneca
  Interventions: Drug: Metoprolol Succinate

INTERVENTIONS:
Drug: Metoprolol Succinate
  Other Names: TOPROL-XL®

SUMMARY:
The purpose of this study is to monitor adverse events, safety and tolerance Metoprolol Succinate Extended-Release Tablets 50 mg under fasting conditions

DETAILED DESCRIPTION:
An open label, balanced, randomized, two-treatment, two-period, two sequence, single dose, crossover, oral bioequivalence study of Metoprolol Succinate Extended-Release tablets 50 mg of Dr. Reddy's Laboratories Limited,under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

Subjects were selected based on the following inclusion criteria:

* Provide written informed consent.
* Must be healthy, adult, human beings between 18 and 45 years of age(both inclusive) weighing at least 50 kg.
* Having a body mass index between 18.5 and 24.9 (both inclusive),calculated as weight in Kg/height in m2
* Must be of normal health as determined by medical history, physical examination and laboratory investigation performed within 28 days prior to the commencement of the study.(Laboratory values must be within normal limits or considered by the physician/investigator to be of no clinical significance).
* Female Subjects of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator (s),such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence.
* surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject)

Exclusion Criteria:

The subjects were excluded based on the following criteria during screening and during the study:

* Incapable of understanding the informed consent.
* Systolic blood pressure less than 90 mm of Hg or more than 140 mm of Hg.
* Diastolic blood pressure less than 60 mm of Hg or more than 90 mm of Hg.
* Oral temperature is below 95.0°F or above 98.6°F.
* Pulse rate below 50/min or above 100/min.
* History of hypersensitivity or idiosyncratic reaction to investigational drug product or any other related drugs.
* Any evidence of impairment of renal, hepatic, cardiac, lung or gastrointestinal function.
* Consumption of grapefruit for the past ten days prior to the check-in, in each period.
* Habit of tobacco chewing.
* Habit of alcoholism and difficulty in abstaining from alcohol during the sample collection period.
* Regular smoker who has a habit of smoking more than nine cigarettes per day and has difficulty in abstaining from smoking during sample collection period.
* Difficulty in abstaining from xanthine containing food or beverages (like tea, coffee, chocolates and cola drinks) during the sample collection period.
* Intake of over the counter (OTC) or prescribed medications and enzyme modifying medication or systemic medication for the last 30 days before dosing.
* Clinically significant abnormalities and lor with significant diseases.
* Confirmed positive in alcohol screening.
* Confirmed positive in selected drug of abuse.
* Participated in any other clinical investigation using experimental drug/donated blood in past 90 days before the date of start of study.
* Confirmed positive in urine pregnancy test.
* Female detected to be pregnant, breast feeding or who is likely to become pregnant during the study.

Ages: 18 Years to 45 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Area under curve (AUC) | Pre-dose (0.00) and 1.00, 2.00, 3.00, 4.00, 5.00, 6.00, 7.00, 8.00, 9.00, 10.00, 11.00, 12.00, 13.00, 14.00, 15.00, 16.00, 18.00, 20.00, 24.00, 36.00 and 48.00 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. P. Vijaya Lakshmi, Clinical Investigator, Principal Investigator — Bioserve Clinical Research Private Limited
Locations (1):
- Bioserve Clinical Research Private Limited, Hyderabad, Andhra Pradesh, India